CLINICAL TRIAL: NCT01669616
Title: Point of Service Diabetes Screening Evaluation
Acronym: POSSE
Status: Completed | Type: Observational
Sponsor: VeraLight, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: VL-2723
Record Dates: First submitted 2012-07-23; First posted 2012-08-21 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Diabetes Mellitus, Non-Insulin Dependent
Keywords: Type 2 Diabetes; Adults 18 years and older
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of the trial is to collect SCOUT DS, random capillary glucose and Hemoglobin A1c measurements from subject 18 years of age or older.

DETAILED DESCRIPTION:
The objectives of this study are to compare the accuracy of SCOUT versus random capillary glucose and several diabetes risk assessment questionnaires for detection of HbA1C-defined dysglycemia.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older

Exclusion Criteria:

* Known to be pregnant (self-reported)
* Receiving dialysis or known renal compromise
* Known to have photosensitivity
* Taking medications that fluoresce
* Have scars, any tattoos, rashes or other disruption/discoloration on the left volar forearm

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Attendees of Blue Cross Blue Shield Wellness Event
Sampling Method: Non-Probability Sample
Enrollment: 667 (Actual)
Dates: Start 2012-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
To compare the accuracy of SCOUT DS versus random capillary glucose and several diabetes risk assessment questionnaires for detection of HbA1c-defined dysglycemia. | one week

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Barrack, MD, Principal Investigator — Blue Cross Blue Shield of Louisiana
Locations (1):
- Blue Cross Blue Shield of Louisiana, Baton Rouge, Louisiana, United States